CLINICAL TRIAL: NCT05278481
Title: Latinos Kick Buts: Mobile Engagement and Cessation Support for Latino Smokers Pilot Study
Brief Title: Latinos Kick Buts: Mobile Engagement and Cessation Support for Latino Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Paula Cupertino, Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: STUDY00006544; R42MD010318 (NIH)
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: 3 x 2 factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Reward Message with standard introduction (Active Comparator)
  Interventions: Behavioral: Reward Message with standard introduction
- Reward Message with culturally tailored introduction (Active Comparator)
  Interventions: Behavioral: Reward Message with culturally tailored introduction
- Threat/Self-efficacy with standard introduction (Active Comparator)
  Interventions: Behavioral: Threat/Self-efficacy with standard introduction
- Threat/Self-efficacy with culturally tailored introduction (Active Comparator)
  Interventions: Behavioral: Threat/Self-efficacy with culturally tailored introduction
- Social norms message with standard introduction (Active Comparator)
  Interventions: Behavioral: Social norms message with standard introduction
- Social norms message with culturally tailored introduction (Active Comparator)
  Interventions: Behavioral: Social norms message with culturally tailored introduction

INTERVENTIONS:
Behavioral: Reward Message with standard introduction — Each text message will be sent 6 times total over two weeks. Each message type will be combined with a standard introduction.
  Arms: Reward Message with standard introduction
Behavioral: Reward Message with culturally tailored introduction — Each text message will be sent 6 times total over two weeks. Each message type will be combined with an introduction culturally tailored for Hispanic/Latino participants.
  Arms: Reward Message with culturally tailored introduction
Behavioral: Threat/Self-efficacy with standard introduction — Each text message will be sent 6 times total over two weeks. Each message type will be combined with a standard introduction.
  Arms: Threat/Self-efficacy with standard introduction
Behavioral: Threat/Self-efficacy with culturally tailored introduction — Each text message will be sent 6 times total over two weeks. Each message type will be combined with an introduction culturally tailored for Hispanic/Latino participants.
  Arms: Threat/Self-efficacy with culturally tailored introduction
Behavioral: Social norms message with standard introduction — Each text message will be sent 6 times total over two weeks. Each message type will be combined with a standard introduction.
  Arms: Social norms message with standard introduction
Behavioral: Social norms message with culturally tailored introduction — Each text message will be sent 6 times total over two weeks. Each message type will be combined with an introduction culturally tailored for Hispanic/Latino participants.
  Arms: Social norms message with culturally tailored introduction

SUMMARY:
Latino Kick Buts (LKB) is a smoking cessation treatment program available to patients identified as smokers at the University of Rochester Medical Center. Latino Kick Buts smoking cessation mobile program encompasses two integrated components: (1) a 12-week text messaging counseling program with interactive capabilities; and (2) pharmacotherapy support (provision of nicotine replacement therapy at no cost). LKB utilization among Latino smokers remains minimal. The aim of this pilot study is to identify types of text message that are more effective to enrolling Latino smokers in the LKB.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Hispanic/Latinos
* be 21 years old or older
* have smoking status recorded in the EMR
* patient of URMedicine

Exclusion Criteria:

* Not Hispanic/Latino
* under 21 years of age
* not a smoker

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Number of participants who enroll in smoking cessation treatment | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No